CLINICAL TRIAL: NCT04574518
Title: Teachable Moment to Opt-out of Tobacco (TeaM OUT): A Stepped Wedge Cluster Randomized Intervention
Brief Title: Teachable Moment to Opt-out of Tobacco: Interactive Voice Response Quit Line for Veteran Active Smokers With Lung Nodules
Acronym: TeaMOUT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency); Ralph H. Johnson VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 19-425
Record Dates: First submitted 2020-09-03; First posted 2020-10-05 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Solitary Pulmonary Nodule; Multiple Pulmonary Nodules; Tobacco Use
Keywords: tobacco use cessation; smoking; evaluation study
MeSH Terms: conditions — Solitary Pulmonary Nodule; Multiple Pulmonary Nodules; Tobacco Use; Tobacco Use Cessation; Smoking

STUDY DESIGN:
Intervention Model Description: The investigators will use a stepped wedge cluster design to randomize at the clinic level (including both community-based outpatient clinics and the main medical center) at each of the 3 sites. The investigators will first institute Enhanced Usual Care for 6 months at each CBOC/medical center. Using a random number generator, the investigators will divide the CBOCs/medical center in the 3 facilities in 4 steps. The investigators will randomize one CBOC at each site to the intervention (interactive voice response quit line) in the first step. For steps 2-4, the investigators will randomize one third of the remaining CBOCs at each facility per step every 6 months.
Masking Description: Participants will not be informed that the intervention is being implemented in a randomized fashion, but they cannot be blinded to the interventions (letter and IVR) they will receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TeaM OUT Intervention (Experimental): The TeaM OUT Intervention has 2 elements: 1) a letter that a) describes the nodule and the importance of cessation related to the pulmonary nodule (i.e. teachable moment) and b) notification that a Proactive IVR Quit line will initiate contact and 2) call(s) from the Proactive IVR Quit Line which a) offers smoking cessation resources and b) helps connect the patient to those resources.
  Interventions: Behavioral: TeaM OUT Intervention
- Enhanced Usual Care (Other): The Enhanced Usual Care arm also has two elements: 1) a letter that a) describes the nodule without linking it to smoking cessation (i.e. no teachable moment) with b) wording to contact an Optional IVR Quit line if desired and 2) the Optional IVR Quit line which a) offers smoking cessation resources and b) helps connect the patient to those resources.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: TeaM OUT Intervention — The TeaM OUT Intervention has 2 elements: 1) a letter that a) describes the nodule and the importance of cessation related to the pulmonary nodule (i.e. teachable moment) and b) notification that a Proactive IVR Quit line will initiate contact and 2) call(s) from the Proactive IVR Quit Line which a) offers smoking cessation resources and b) helps connect the patient to those resources.
  Arms: TeaM OUT Intervention
Behavioral: Enhanced Usual Care — The Enhanced Usual Care arm also has two elements: 1) a letter that a) describes the nodule without linking it to smoking cessation (i.e. no teachable moment) with b) wording to contact an Optional IVR Quit line if desired and 2) the Optional IVR Quit line which a) offers smoking cessation resources and b) helps connect the patient to those resources.
  Arms: Enhanced Usual Care

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a smoking cessation outreach intervention (TeaM OUT) on increasing use of smoking cessation resources in Veterans. The hypotheses are 1) patients included in the TeaM OUT group will have higher accession of cessation services, such as counseling and medication therapies, compared to patients in enhanced usual care and 2) more patients in the TeaM OUT group will have quit smoking at one year after the intervention.

Veterans with a recently diagnosed lung nodule who currently smoke will receive the TeaM OUT intervention or Enhanced Usual Care. The TeaM OUT intervention has 2 parts: 1) a letter that a) describes the nodule and the importance of cessation related to the pulmonary nodule (i.e. teachable moment) and b) notification that a Proactive IVR Quit Line will initiate contact and 2) call(s) from the Proactive IVR Quit Line which a) offers smoking cessation resources and b) helps connect the patient to those resources. The enhanced usual care group will receive a letter that provides information about how to contact the IVR Quit Line.

The IVR system will track referrals to cessation services. Additional information about smoking status and use of cessation resources will be collected from the electronic health record and surveys.

.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed pulmonary nodule with plan for surveillance
* Active smoker
* Receiving care at the Portland VA Health Care System, the Minneapolis VA Health Care System, or the Ralph H. Johnson Medical Center (Charleston, SC VA)

Exclusion Criteria:

-No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
IVR connection to smoking cessation service | 56 weeks after nodule identification
  A positive (yes) response is a completed call to a patient who then indicates (by pressing the number keypad) to be connected to one or more smoking cessation resources. In the control group, if the patient calls the Optional IVR Quitline and then requests to be connected to smoking cessation resources it is counted as a positive response. Each patient will be categorized as a "yes" after her/his first positive response to the system, regardless of how many times he/she actually engages with the system.
7-day point prevalence nicotine abstinence | 56 weeks after exposure to TeaM OUT Intervention or Enhanced Usual Care
  Aim 2: Participants will be considered to have quit smoking (including non-combustible) if they respond "no" to the question, "Have you smoked a cigarette (regular or e-cigarette), even a puff, in the past 7 days?"

SECONDARY OUTCOMES:
Utilization of cessation resources | 72 weeks after nodule identification
  Aim 1: Utilization includes new prescriptions and refills for nicotine-replacement therapies, anti-smoking medications, referrals to smoking cessation counseling, and attendance of smoking cessation counseling session, as recorded in the electronic health record.
Incremental Behavior Change Toward Smoking Cessation (IBC-S) | 56 weeks after exposure to TeaM OUT Intervention or Enhanced Usual Care
  Aim 2: Measure is the summed score of the Incremental Behavior Change toward Smoking cessation (IBC-S) scale.

OTHER OUTCOMES:
Qualitative analysis of IVR intervention | Patients--56 weeks after exposure to TeaM OUT Intervention or Enhanced Usual Care; Clinical Stakeholders--at least 6 months after clinic randomization
  Aim 3: Interviews with patients and clinical stakeholders will collect feedback about the IVR intervention. Interview content will be analyzed using qualitative description. Interview transcripts will be reviewed and coded by the qualitative analysts. Development of the codes will occur in the context of the qualitative data. The analysts will discuss the codes, achieve consensus, resolve differences, and modify the codes if necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher G. Slatore, MD MS, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (3):
- United States (3):
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be saved in our IRB-approved Health Services Research Repository (Portland VA IRB #3535) at the conclusion of the study and requests for access can be submitted to the study team.
Time Frame: Conclusion of the study, estimated to be January 2027

REFERENCES:
- [Background] Reinke LF, Sullivan DR, Slatore C, Dransfield MT, Ruedebusch S, Smith P, Rise PJ, Tartaglione EV, Vig EK, Au DH. A Randomized Trial of a Nurse-Led Palliative Care Intervention for Patients with Newly Diagnosed Lung Cancer. J Palliat Med. 2022 Nov;25(11):1668-1676. doi: 10.1089/jpm.2022.0008. Epub 2022 Jun 1. PMID 35649214
- [Background] Wiener RS, Barker AM, Carter-Harris L, Caverly TJ, Crocker DA, Denietolis A, Doherty C, Fagerlin A, Gallagher-Seaman M, Gould MK, Han PKJ, Herbst AN, Ito Fukunaga M, McCullough MB, Miano DA, Quaife SL, Slatore CG, Fix GM. Stakeholder Research Priorities to Promote Implementation of Shared Decision-Making for Lung Cancer Screening: An American Thoracic Society and Veterans Affairs Health Services Research and Development Statement. Am J Respir Crit Care Med. 2022 Mar 15;205(6):619-630. doi: 10.1164/rccm.202201-0126ST. PMID 35289730
- [Background] Nunez ER, Caverly TJ, Zhang S, Glickman ME, Qian SX, Boudreau JH, Miller DR, Slatore CG, Wiener RS. Factors Associated With Declining Lung Cancer Screening After Discussion With a Physician in a Cohort of US Veterans. JAMA Netw Open. 2022 Aug 1;5(8):e2227126. doi: 10.1001/jamanetworkopen.2022.27126. PMID 35972738
- [Background] Lewis JA, Wiener RS, Slatore CG, Spalluto LB. Doing Versus Documenting Shared Decision-Making for Lung Cancer Screening-Are They the Same? J Am Coll Radiol. 2022 Aug;19(8):954-956. doi: 10.1016/j.jacr.2022.03.019. Epub 2022 May 18. No abstract available. PMID 35594952
- [Background] Slatore CG, Golden SE, Thomas T, Patzel M, Bumatay S, Shannon J, Davis M. Beliefs and Practices of Primary Care Providers Regarding Performing Low-Dose CT Studies for Lung Cancer Screening. Chest. 2022 Mar;161(3):853-859. doi: 10.1016/j.chest.2021.08.062. Epub 2021 Sep 1. No abstract available. PMID 34480957
- [Background] Lewis JA, Samuels LR, Denton J, Matheny ME, Maiga A, Slatore CG, Grogan E, Kim J, Sherrier RH, Dittus RS, Massion PP, Keohane L, Roumie CL, Nikpay S. The Association of Health Care System Resources With Lung Cancer Screening Implementation: A Cohort Study. Chest. 2022 Sep;162(3):701-711. doi: 10.1016/j.chest.2022.03.050. Epub 2022 Apr 9. PMID 35413280
- [Background] Braithwaite D, Karanth SD, Slatore CG, Zhang D, Bian J, Meza R, Jeon J, Tammemagi M, Schabath M, Wheeler M, Guo Y, Hochhegger B, Kaye FJ, Silvestri GA, Gould MK. Personalised Lung Cancer Screening (PLuS) study to assess the importance of coexisting chronic conditions to clinical practice and policy: protocol for a multicentre observational study. BMJ Open. 2022 Jun 22;12(6):e064142. doi: 10.1136/bmjopen-2022-064142. PMID 35732383
- [Background] Wang Q, Stone K, Kern JA, Slatore CG, Swanson S, Blackstock W Jr, Khan RS, Smith CB, Veluswamy RR, Chidel M, Wisnivesky JP. Adverse Events Following Limited Resection versus Stereotactic Body Radiation Therapy for Early Stage Lung Cancer. Ann Am Thorac Soc. 2022 Dec;19(12):2053-2061. doi: 10.1513/AnnalsATS.202203-275OC. PMID 35816617
- [Background] Gundle K, Hooker ER, Golden SE, Shull S, Crothers K, Melzer AC, Slatore CG. Use of Veterans Health Administration Structured Data to Identify Patients Eligible for Lung Cancer Screening. Mil Med. 2023 Jul 22;188(7-8):e2419-e2423. doi: 10.1093/milmed/usad017. PMID 36722178
- [Background] Golden SE, Schweiger L, Melzer AC, Ono SS, Datta S, Davis JM, Slatore CG. "It's a decision I have to make": Patient perspectives on smoking and cessation after lung cancer screening decisions. Prev Med Rep. 2022 Oct 5;30:102014. doi: 10.1016/j.pmedr.2022.102014. eCollection 2022 Dec. PMID 36237837
- [Background] Nunez ER, Slatore CG, Tanner NT, Melzer AC, Crothers KA, Lewis JA, Fabbrini AE, Brown JK, Wiener RS. National Survey of Lung Cancer Screening Practices in Veterans Health Administration Facilities. Am J Prev Med. 2023 Nov;65(5):901-905. doi: 10.1016/j.amepre.2023.05.005. Epub 2023 May 9. PMID 37169315
- [Background] Kearney LE, Butler C, Nunez ER, Qian S, Slatore CG, Spalluto L, Wiener RS. Highly variable reporting of incidental findings in a national cohort of US veterans screened for lung cancer. Clin Imaging. 2023 Aug;100:21-23. doi: 10.1016/j.clinimag.2023.04.017. Epub 2023 May 2. No abstract available. PMID 37146522
- [Background] Nugent SM, Slatore CG, Winchell K, Handley R, Clayburgh D, Chandra R, Hooker ER, Knight SJ, Morasco BJ. Prevalence and correlates of high-dose opioid use among survivors of head and neck cancer. Head Neck. 2023 Aug;45(8):2058-2067. doi: 10.1002/hed.27432. Epub 2023 Jun 27. PMID 37366072
- [Background] Vranas KC, Hooker ER, Golden SE, Nugent S, Slatore CG. Association of Communication Quality With Patient-Centered Outcomes Among Patients With Incidental Pulmonary Nodules. Chest. 2023 Aug;164(2):556-559. doi: 10.1016/j.chest.2023.03.009. Epub 2023 Mar 11. No abstract available. PMID 36907374
- [Background] Rozema EJ, Creekmur B, Musigdilok VV, Steltz J, Gould MK, Slatore CG. Patient responses to passive enrollment into a large, pragmatic clinical trial: A qualitative content analysis. Contemp Clin Trials. 2022 Oct;121:106925. doi: 10.1016/j.cct.2022.106925. Epub 2022 Sep 13. PMID 36108887
- [Background] Gogebakan KC, Lange J, Slatore CG, Etzioni R. Modeling the impact of novel systemic treatments on lung cancer screening benefits. Cancer. 2023 Jan 15;129(2):226-234. doi: 10.1002/cncr.34527. Epub 2022 Nov 1. PMID 36320180
- [Background] Rustagi AS, Byers AL, Brown JK, Purcell N, Slatore CG, Keyhani S. Lung Cancer Screening Among U.S. Military Veterans by Health Status and Race and Ethnicity, 2017-2020: A Cross-Sectional Population-Based Study. AJPM Focus. 2023 Feb 9;2(2):100084. doi: 10.1016/j.focus.2023.100084. eCollection 2023 Jun. PMID 37790642
- [Background] Sullivan DR, Vranas KC, Delorit M, Golden SE, Slatore CG, Ganzini L, Hansen L. Relationships among clinicians are crucial to successful palliative care integration: a qualitative study in lung cancer. Future Oncol. 2023 Jan;19(3):245-257. doi: 10.2217/fon-2022-0958. Epub 2023 Mar 28. PMID 36974605
- [Background] Sullivan DR, Wisnivesky JP, Nugent SM, Stone K, Farris MK, Kern JA, Swanson S, Smith CB, Rosenzweig K, Slatore CG. Decision Regret among Patients with Early-stage Lung Cancer Undergoing Radiation Therapy or Surgical Resection. Clin Oncol (R Coll Radiol). 2023 Jun;35(6):e352-e361. doi: 10.1016/j.clon.2023.03.015. Epub 2023 Mar 29. PMID 37031075
- [Background] Golden SE, Disher N, Dieckmann NF, Eden KB, Matlock D, Vranas KC, Slatore CG, Sullivan DR. Show me the roads and give me a road map: Development of a patient conversation tool to improve lung cancer treatment decision-making. PEC Innov. 2022 Oct 21;1:100094. doi: 10.1016/j.pecinn.2022.100094. eCollection 2022 Dec. PMID 37213736
- [Background] Lewis JA, Samuels LR, Weems J, Park D, Winter R, Lindsell CJ, Callaway-Lane C, Audet C, Slatore CG, Wiener RS, Dittus RS, Kripalani S, Yankelevitz DF, Henschke CI, Moghanaki D, Matheny ME, Vogus TJ, Roumie CL, Spalluto LB. The Association of Organizational Readiness With Lung Cancer Screening Utilization. Am J Prev Med. 2023 Nov;65(5):844-853. doi: 10.1016/j.amepre.2023.05.018. Epub 2023 May 22. PMID 37224985
- [Background] Hooker ER, Chapa J, Vranas KC, Niederhausen M, Goodlin SJ, Slatore CG, Sullivan DR. Intersection of Palliative Care and Hospice Use Among Patients With Advanced Lung Cancer. J Palliat Med. 2023 Nov;26(11):1474-1481. doi: 10.1089/jpm.2023.0040. Epub 2023 Jun 1. PMID 37262128
- [Background] Gould MK, Creekmur B, Qi L, Golden SE, Kaplan CP, Walter E, Mularski RA, Vaszar LT, Fennig K, Steiner J, de Bie E, Musigdilok VV, Altman DA, Dyer DS, Kelly K, Miglioretti DL, Wiener RS, Slatore CG, Smith-Bindman R. Emotional Distress, Anxiety, and General Health Status in Patients With Newly Identified Small Pulmonary Nodules: Results From the Watch the Spot Trial. Chest. 2023 Dec;164(6):1560-1571. doi: 10.1016/j.chest.2023.06.022. Epub 2023 Jun 24. PMID 37356710
- [Background] Rustagi AS, Slatore CG, Keyhani S. Self-Rated Health and Ability to Climb Stairs: A Pragmatic Health Assessment Before Lung Cancer Screening. Ann Intern Med. 2023 Apr;176(4):568-571. doi: 10.7326/M22-3598. Epub 2023 Mar 7. No abstract available. PMID 36877963
- [Result] Unger S, Golden SE, Melzer AC, Tanner N, Deepak J, Delorit M, Scott JY, Slatore CG. Study design for a proactive teachable moment tobacco treatment intervention among patients with pulmonary nodules. Contemp Clin Trials. 2022 Oct;121:106908. doi: 10.1016/j.cct.2022.106908. Epub 2022 Sep 8. PMID 36087843
- [Result] Golden SE, Unger S, Slatore CG. Implementing Smoking Cessation Telehealth Technologies Within the VHA: Lessons Learned. Fed Pract. 2023 Aug;40(8):256-260. doi: 10.12788/fp.0393. Epub 2023 Aug 11. PMID 37868257

DOCUMENTS (1):
  • Informed Consent Form (2022-11-03): https://cdn.clinicaltrials.gov/large-docs/18/NCT04574518/ICF_000.pdf